CLINICAL TRIAL: NCT05425017
Title: Simultaneous Crepitus and Diagnostic Ultrasound Assessment of the Lumbar Zygapophyseal Joints Expansion of Validation and Reliability of Automated Analysis of Crepitus in Human Subjects
Brief Title: Analysis of Crepitus in Human Subjects
Acronym: CrUS
Status: Active, not recruiting | Type: Observational
Sponsor: National University of Health Sciences (Other)
Collaborators: Yale University (Other)
Responsible Party: Principal Investigator, Gregory D. Cramer, Professor and Dean of Research, National University of Health Sciences
Other Study IDs: H2101/H2302
Record Dates: First submitted 2022-06-15; First posted 2022-06-21 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-11

CONDITIONS: Low Back Pain; Healthy
Keywords: crepitus; spine; noise; physiological; pathological
MeSH Terms: conditions — Low Back Pain | interventions — Range of Motion, Articular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Low back pain group: Participants currently experiencing low back pain will have small accelerometers taped along spine, Ultrasound (US) Clinician will place an US transducer at the right L4/L5 Z joint. Participants will complete a range of motions while accelerometers are recording back sounds. Subsequently, they will receive a chiropractic adjustment, then repeat the range of motions
  Interventions: Other: Range of motion with spinal adjustment
- Healthy group: Participants without low back pain will have small accelerometers taped along spine. Ultrasound (US) Clinician will place a US transducer at the right L4/L5 Z joint. Participants will perform a range of motions while accelerometers are recording back sounds. Subsequently, they will receive a chiropractic adjustment, then repeat the range of motions
  Interventions: Other: Range of motion with spinal adjustment

INTERVENTIONS:
Other: Range of motion with spinal adjustment — With accelerometers affixed to spine recording vibrations, the participants complete range of motion. After completing, they receive a low back spinal adjustment and repeat range of motion

SUMMARY:
Chiropractic adjustment has been shown to gap certain joints in the spine, thereby improving mobility in individuals with decreased movement capabilities. During normal motion, joints in the spine produce sounds and vibrations called crepitus. The purpose of this study is to assess how this crepitus may be used as an indicator for joint degeneration in healthy human subjects and those with low back pain, and if chiropractic adjusting causes change in this crepitus. The investigators hypothesize that change in crepitus after adjustment may be a useful indication of changes in joint mobility and joint stiffness.

DETAILED DESCRIPTION:
Objective: This is an expansion of the initial study "Analysis of Crepitus in Human Subjects" to assess the feasibility of simultaneously recording zygapophyseal (Z) joint crepitus using piezoelectric accelerometers and Z joint motion using diagnostic ultrasound (US), and qualitatively assess the US images with particular focus on images taken of Z joints exhibiting crepitus. Like the original study (n=12), the results of a recently developed automated method (AM) is compared with two human observers in the analysis of recordings of human lumbar zygapophyseal (Z) joint crepitus. The recordings will be taken during ranges of motion performed before and after lumbar side-posture spinal manipulation (SMT). Methods: Six (6) healthy and 6 low back pain subjects will participate in the study. Using clinical study procedures developed previously, subjects will be given an initial phone screen before being scheduled for a clinical study appointment. At the appointment, subjects will undergo the informed consent process, and those consenting will be further screened and examined by the Research Clinician who will use the inclusion/exclusion criteria to determine eligibility for the study. Eligible subjects will be enrolled and scheduled for an accelerometry visit. At the accelerometry visit, 11 accelerometers will be applied to the lumbar region, allowing assessment of Z joint crepitus. US imaging of the right L4/L5 Z joint will be included. Each subject will undergo full flexion and full extension (ROM) while recordings are made from the accelerometers. Subjects will then undergo bilateral lumbar SMT, and immediately thereafter will undergo repeated ROM while recordings are made. Two human observers and the AM, blinded to the results of one another, will then assess the recordings to identify Z joints from which crepitus originated. The primary outcomes will be: 1) weighted kappa inter-rater reliability statistic comparing AM and the 2 human observers in identifying Z joint crepitus, and 2) ANOVA test statistic comparing time to complete the crepitus analysis by the AM and human observers. Hypotheses: 1) The automated method will be reliable, agreeing with the human observers' analysis. 2) The automated method will be significantly more time efficient than the analyses made by the human observers. Application: The investigators believe that this program will improve the efficiency of identifying the site of Z joint crepitus, thereby advancing the line of investigation designed to use crepitus as a biomarker of spinal joint dysfunction.

ELIGIBILITY:
Inclusion Criteria:

Healthy (no LBP) Subjects (n=6):

* 30 to 75 years of age
* No previous history of LBP lasting for more than two weeks, or no more than three episodes of back pain of brief duration (one week) in any given year (to recruit healthy subjects with no history, or a minimal history, of LBP).
* No presence of current LBP
* Female with a BMI of 28 or less; Male with a BMI of 30 or less.

LBP Subjects Criteria (n=6):

* 30 to 75 years of age
* Current LBP of at least one-week (7 days) duration
* Female with a BMI of 28 or less; Male with a BMI of 30 or less.

Exclusion Criteria:

Healthy Subjects:

* Under 30 or over 75 years of age
* History of an episode of LBP lasting for more than two weeks, or more than three episodes of back pain of brief duration (one week) in any given year (see reasons for no LBP in Inclusion Criteria)
* Presence of Current LBP
* Prior spinal surgery
* Presence of current spinal fracture, tumor, infection, or scoliosis of greater than 5 degrees (Cobb's angle, scoliosis decreases ability to place the accelerometers); or other known significant pathology
* Known allergies to latex or adhesives (including Band-Aids) applied to the skin (accelerometers are taped to the skin)
* BMI over 30 for males; BMI over 28 for females (subject will be weighed at exam)
* Pregnancy (because of unique biomechanical patterns and changes in the ranges of motion that occur during pregnancy)
* Positive findings on any of the orthopedic or neurological tests listed on exam form; (because these subjects will be assessed as healthy individuals, indication of somatic pathology or neurological deficit are exclusionary criteria)
* Decreased range of motion (as measured with a goniometer) of the lumbar region (recording during flexion and extension ranges of motion are conducted in the study; consequently a full range of motion is necessary for the healthy subjects). The following ranges will be exclusionary: Flexion: < 40º (normal = 60º); Extension: < 10º (normal = 20º);
* Pain or discomfort during set-up for lumbar side-posture spinal manipulation (SMT) or during lumbar SMT given at the conclusion of the examination (the study assesses changes following SMT, consequently ability to tolerate SMT is important)
* Contraindication to manipulative treatment

LBP Subjects:

* Under 30 or over 75 years of age
* Absence of Current LBP of at least one-week (7 days) duration
* BMI over 30 for males; BMI over 28 for females (subject will be weighed at exam)
* Known allergies to latex or adhesives (including Band Aids) applied to the skin (accelerometers are taped to the skin)
* Pregnancy (because of unique biomechanical patterns and changes in the ranges of motion that occur during pregnancy)
* Pain radiating below the knee
* Presence of current spinal fracture, tumor, infection, or scoliosis of greater than 5 degrees (Cobb's angle, scoliosis decreases ability to place the accelerometers); or other known significant pathology
* Prior spinal surgery
* Negative findings on all of the orthopedic or neurological tests listed on exam form
* Contraindication to manipulative treatment

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from the faculty, student and staff population at National University Of Health Sciences, Lombard, IL. If unable to recruit sufficient number of participants, recruitment will be extended to the general population of the Chicago, IL metro area.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Inter-rater reliability of analysis of spinal crepitus produced during range of motion | 6 month following data collection
  Piezoelectric accelerometers are taped to the participants spine. The participant then completes a range of motions while the accelerometers are recording any sounds being produced during the movement. Following range of motion, the participant receives a side posture chiropractic adjustment and then repeats the range of motion while the accelerometers are recording. All participant recordings will be collected prior to the start of analysis. Utilizing previously validated methods to analyze accelerometer recordings taken during participants range of motion, spinal crepitus will be identified and defined and programmed into a computer automated method of analysis. Kappa inter-rater reliability statistic will be compare consensus of two human observers to the computer automated method of analysis will be compared.
Time of analysis of spinal crepitus produced during range of motion | 6 month following data collection
  Piezoelectric accelerometers are taped to the participants spine. The participant then completes a range of motions while the accelerometers are recording any sounds being produced during the movement. Following range of motion, the participant receives a side posture chiropractic adjustment and then repeats the range of motion while the accelerometers are recording. All participant recordings will be collected prior to the start of analysis. Utilizing previously validated methods to analyze accelerometer recordings taken during participants range of motion, spinal crepitus will be identified and defined and programmed into a computer automated method of analysis. The time it takes to complete analysis of all crepitus recordings will be compared by ANOVA between two human observers and the computer automated method of analysi

SECONDARY OUTCOMES:
Change in crepitus following spinal manipulation | 6 month following data collection
  Piezoelectric accelerometers are taped to the participants spine. The participant then completes a range of motions while the accelerometers are recording any sounds being produced during the movement. Following range of motion, the participant receives a side posture chiropractic adjustment and then repeats the range of motion while the accelerometers are recording. For each participant, crepitus produced during range of motion performed prior to chiropractic adjustment will be compared to crepitus produced following chiropractic adjustment. All participant recordings will be collected prior to the start of analysis. Ultrasound outcomes will be subjective and descriptive to identify imaging of the right L4/L5 Z joint.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Cramer, DC, PhD, Principal Investigator — National University of Health Sciences; Gregory Roytman, DC, Principal Investigator — Yale University
Locations (2):
- United States (2):
  - National University of Health Sciences, Lombard, Illinois
  - National University of Health Science, Lombard, Illinois

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hoy D, March L, Brooks P, Blyth F, Woolf A, Bain C, Williams G, Smith E, Vos T, Barendregt J, Murray C, Burstein R, Buchbinder R. The global burden of low back pain: estimates from the Global Burden of Disease 2010 study. Ann Rheum Dis. 2014 Jun;73(6):968-74. doi: 10.1136/annrheumdis-2013-204428. Epub 2014 Mar 24. PMID 24665116
- [Background] Bronfort G, Haas M, Evans RL, Bouter LM. Efficacy of spinal manipulation and mobilization for low back pain and neck pain: a systematic review and best evidence synthesis. Spine J. 2004 May-Jun;4(3):335-56. doi: 10.1016/j.spinee.2003.06.002. PMID 15125860
- [Background] Chou R, Huffman LH; American Pain Society; American College of Physicians. Nonpharmacologic therapies for acute and chronic low back pain: a review of the evidence for an American Pain Society/American College of Physicians clinical practice guideline. Ann Intern Med. 2007 Oct 2;147(7):492-504. doi: 10.7326/0003-4819-147-7-200710020-00007. PMID 17909210
- [Background] Schneider M, Haas M, Glick R, Stevans J, Landsittel D. Comparison of spinal manipulation methods and usual medical care for acute and subacute low back pain: a randomized clinical trial. Spine (Phila Pa 1976). 2015 Feb 15;40(4):209-17. doi: 10.1097/BRS.0000000000000724. PMID 25423308
- [Background] Fritz JM, Kim J, Dorius J. Importance of the type of provider seen to begin health care for a new episode low back pain: associations with future utilization and costs. J Eval Clin Pract. 2016 Apr;22(2):247-52. doi: 10.1111/jep.12464. Epub 2015 Sep 29. PMID 26417660
- [Background] Deyo RA, Dworkin SF, Amtmann D, Andersson G, Borenstein D, Carragee E, Carrino J, Chou R, Cook K, DeLitto A, Goertz C, Khalsa P, Loeser J, Mackey S, Panagis J, Rainville J, Tosteson T, Turk D, Von Korff M, Weiner DK. Report of the NIH Task Force on Research Standards for Chronic Low Back Pain. Int J Ther Massage Bodywork. 2015 Sep 1;8(3):16-33. doi: 10.3822/ijtmb.v8i3.295. eCollection 2015 Sep. PMID 26388962
- [Background] Rubinstein SM, Terwee CB, Assendelft WJ, de Boer MR, van Tulder MW. Spinal manipulative therapy for acute low-back pain. Cochrane Database Syst Rev. 2012 Sep 12;2012(9):CD008880. doi: 10.1002/14651858.CD008880.pub2. PMID 22972127
- [Background] Deyo RA, Bryan M, Comstock BA, Turner JA, Heagerty P, Friedly J, Avins AL, Nedeljkovic SS, Nerenz DR, Jarvik JG. Trajectories of symptoms and function in older adults with low back disorders. Spine (Phila Pa 1976). 2015 Sep 1;40(17):1352-62. doi: 10.1097/BRS.0000000000000975. PMID 25996537
- [Background] Brennan GP, Fritz JM, Hunter SJ, Thackeray A, Delitto A, Erhard RE. Identifying subgroups of patients with acute/subacute "nonspecific" low back pain: results of a randomized clinical trial. Spine (Phila Pa 1976). 2006 Mar 15;31(6):623-31. doi: 10.1097/01.brs.0000202807.72292.a8. PMID 16540864
- [Background] Cramer GD, Ross JK, Raju PK, Cambron JA, Dexheimer JM, Bora P, McKinnis R, Selby S, Habeck AR. Distribution of cavitations as identified with accelerometry during lumbar spinal manipulation. J Manipulative Physiol Ther. 2011 Nov;34(9):572-83. doi: 10.1016/j.jmpt.2011.05.015. Epub 2011 Jul 18. PMID 21986305
- [Background] Cramer GD, Ross K, Pocius J, Cantu JA, Laptook E, Fergus M, Gregerson D, Selby S, Raju PK. Evaluating the relationship among cavitation, zygapophyseal joint gapping, and spinal manipulation: an exploratory case series. J Manipulative Physiol Ther. 2011 Jan;34(1):2-14. doi: 10.1016/j.jmpt.2010.11.008. PMID 21237402
- [Background] Cramer GD, Budavich M, Bora P, Ross K. A Feasibility Study to Assess Vibration and Sound From Zygapophyseal Joints During Motion Before and After Spinal Manipulation. J Manipulative Physiol Ther. 2017 Mar-Apr;40(3):187-200. doi: 10.1016/j.jmpt.2017.01.003. Epub 2017 Mar 6. PMID 28268027
- [Background] Cramer GD, Ross K, Raju PK, Cambron J, Cantu JA, Bora P, Dexheimer JM, McKinnis R, Habeck AR, Selby S, Pocius JD, Gregerson D. Quantification of cavitation and gapping of lumbar zygapophyseal joints during spinal manipulative therapy. J Manipulative Physiol Ther. 2012 Oct;35(8):614-21. doi: 10.1016/j.jmpt.2012.06.007. Epub 2012 Aug 14. PMID 22902194
- [Background] Lascelles BD, Dong YH, Marcellin-Little DJ, Thomson A, Wheeler S, Correa M. Relationship of orthopedic examination, goniometric measurements, and radiographic signs of degenerative joint disease in cats. BMC Vet Res. 2012 Jan 27;8:10. doi: 10.1186/1746-6148-8-10. PMID 22281125
- [Background] Abhishek A, Doherty M. Diagnosis and clinical presentation of osteoarthritis. Rheum Dis Clin North Am. 2013 Feb;39(1):45-66. doi: 10.1016/j.rdc.2012.10.007. PMID 23312410
- [Background] Robertson CJ. Joint crepitus--are we failing our patients? Physiother Res Int. 2010 Dec;15(4):185-8. doi: 10.1002/pri.492. Epub 2010 Oct 28. No abstract available. PMID 21031637
- [Background] Henderson CN, Cramer GD, Zhang Q, DeVocht JW, Fournier JT. Introducing the external link model for studying spine fixation and misalignment: part 2, Biomechanical features. J Manipulative Physiol Ther. 2007 May;30(4):279-94. doi: 10.1016/j.jmpt.2007.03.002. PMID 17509437
- [Background] Cramer GD, Henderson CN, Little JW, Daley C, Grieve TJ. Zygapophyseal joint adhesions after induced hypomobility. J Manipulative Physiol Ther. 2010 Sep;33(7):508-18. doi: 10.1016/j.jmpt.2010.08.002. PMID 20937429
- [Result] Roytman G, Faydenko J, Budavich M, Pocius JD, Cramer G. Automated Vibration and Acoustic Crepitus Sensing in Humans. J. Tribol. Sept 2023, 145 (9)